CLINICAL TRIAL: NCT03763643
Title: PRI-VENT FSGS: Preemptive Rituximab to Prevent Recurrent Focal Segmental Glomerulosclerosis Post-Transplant
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: University of Minnesota (Other)
Collaborators: United States Department of Defense (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: PEDS-2018-25868
Record Dates: First submitted 2018-08-07; First posted 2018-12-04 (Actual); Last update posted 2025-09-10 (Actual); Status verified 2025-09

CONDITIONS: Focal Segmental Glomerulosclerosis
MeSH Terms: conditions — Glomerulosclerosis, Focal Segmental | interventions — Rituximab; Plasmapheresis

STUDY DESIGN:
Intervention Model Description: Control group and treatment/intervention group. Pilot/feasibility study.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Rituximab + plasmapharesis (Experimental): This is a phase III, multicenter, randomized, open-label clinical trial. Participants with FSGS will be randomized 1:1 to receive rituximab or placebo on day -1, 0 and +1 prior to or after kidney transplantation in addition to standard plasmapheresis.
  Interventions: Drug: Rituximab; Procedure: Plasmapheresis
- Placebo + plasmapharesis (Placebo Comparator): This is a phase III, multicenter, randomized, open-label clinical trial. Participants with FSGS will be randomized 1:1 to receive rituximab or placebo on day -1, 0 and +1 prior to or after kidney transplantation in addition to standard plasmapheresis.
  Interventions: Procedure: Plasmapheresis

INTERVENTIONS:
Drug: Rituximab — Rituximab 375mg/m2 intravenous on day 0 or -1 prior to kidney transplant
  Arms: Rituximab + plasmapharesis
Procedure: Plasmapheresis — 1.5 volume exchange plasmapheresis with fresh frozen plasma replacement

SUMMARY:
This is a pilot/feasibility, multicenter, randomized, open label, clinical trial to test that hypothesis that plasmapheresis plus rituximab prior to or at the time of kidney transplantation can prevent recurrent FSGS in children and adults.

DETAILED DESCRIPTION:
Recurrent FSGS is a risk factor for graft lost: Recurrence of FSGS can occur rapidly, within minutes of transplantation, and can lead to immediate onset of proteinuria and graft dysfunction. Recurrent FSGS is definitively diagnosed with a kidney biopsy. Early kidney biopsies in recurrent FSGS often demonstrate only extensive foot process effacement with the classic focal sclerosis appearing only after months of proteinuria. Recurrent FSGS is the single most important cause of graft failure in patients with FSGS. Patients with recurrent FSGS have significantly decreased graft survival compared to patients without recurrence and often require multiple kidney transplants in their lifetime. A number of clinical risk factors for recurrent FSGS have been identified including prior recurrence, Caucasian race, rapid progression of primary FSGS to ESRD within 3 years, mesangial hypercellularity on primary biopsy and living donor transplant, however these findings are inconsistent among various small studies. 3 A recent study from Europe identified late steroid resistant FSGS (nephrotic syndrome that is initially responsive to steroids, then later resistant) as a strong risk factor for recurrence. These findings have been replicated in our recent retrospective study of a North American cohort from the Midwest Pediatric Nephrology Consortium (N=116) that showed risk of recurrent FSGS was 70.6% in children with late steroid resistant FSGS compared to 35.8% risk in children with initial steroid resistant FSGS (manuscript in preparation). Genetic risk factors for late steroid resistant FSGS are unknown. In the same study Investigators identified native kidney biopsy findings that may predict risk of recurrence. Unfortunately, an individual's risk of recurrent disease cannot be predicted accurately prior to transplant. Thus, patients with FSGS have a high risk of recurrent disease post-transplant that is difficult to predict and patients have poor kidney transplant outcomes.

Plasmapheresis is utilized as a treatment for recurrent FSGS once it occurs: Several therapies for recurrent FSGS have been attempted with varying degrees of success but there remains no proven treatment for recurrent FSGS post-transplant. 7-10 The demonstration of a possible causative circulating factor by Savin et. al. 11 galvanized the field to attempt plasmapheresis to remove 'the permeability factor' as a therapy for recurrent FSGS. Therefore, recurrent FSGS is most often treated with plasmapheresis to remove the circulating factor and this is effective in a subset of patients. The results of uncontrolled single center case reports and series suggest a benefit from plasmapheresis 12-14 although graft loss from recurrent disease remains unacceptably high. Patients who do not respond to plasmapheresis have rapidly progressive chronic kidney disease. These patients have been treated with alternate agents such as rituximab, abatacept, or high dose cyclosporine with variable responses.15-17 Ideally, therapies will be identified to prevent recurrent FSGS before it occurs. Prevention of recurrent FSGS will lead to longer kidney transplant survival and reduced health care costs.

No treatments are available to prevent the recurrence of FSGS after transplant: Since 2005, there have been 3 published studies that have utilized a variety of protocols of plasmapheresis for the prevention of recurrent FSGS with inconsistent results. 18-20 The University of Minnesota pediatric transplant program has utilized pre-emptive plasmapheresis in children at risk for recurrent FSGS since 2006. In a recent review of our data, the incidence of recurrent FSGS post-transplant was not significantly different in patients who had undergone pre-emptive prophylactic plasmapheresis versus historic controls who had not (31% vs. 23%, p 0.5) (manuscript in press). Although this is a retrospective study, the data seems to suggest that plasmapheresis alone is not effective for preventing recurrence of FSGS. In addition, as stated above, the benefit of plasmapheresis in the treatment of recurrence is reported. 12-14 Thus, plasmapheresis with additional preemptive strategies to prevent recurrent FSGS are needed.

Rituximab has been used to treat recurrent FSGS and is a promising novel therapy to prevent recurrent disease. Rituximab is a chimeric monoclonal antibody against CD20 on B cells that leads to B cell depletion that has been used successfully for the treatment of primary steroid sensitive nephrotic syndrome as well as steroid sensitive and resistant FSGS. 21,22 Rituximab may act in FSGS via alterations in B-cell/T-cell interactions leading to changes in cytokine secretion or co-stimulation. Alternately, rituximab may have a direct effect on podocyte structure and function as it has been found to bind directly to the sphingomyelin phosphodiesterase acid-like 3b protein on the surface of podocytes. 23 Recent systematic reviews on the use of rituximab in the treatment of post-transplant FSGS (either with or without plasmapheresis) demonstrate partial or complete remission in ~60% of treated patients.15,24 The use of preemptive rituximab has been reported to be effective in preventing recurrent FSGS in 4 patients at very high risk due to prior graft loss from recurrent disease, however randomized controlled trials have not been performed. 25 Given the effectiveness of rituximab in the treatment of some patients with both primary and recurrent FSGS and the report of successful preemptive use of rituximab in high risk transplant patients, treatment with Rituximab in patients with FSGS prior to kidney transplant is a promising novel therapy to prevent recurrent disease. Preventing recurrent FSGS, rather than treating it once it has already occurred, is likely to minimize graft injury and prolong graft life, therefore preemptive strategies are needed.

ELIGIBILITY:
In order to be eligible to participate in this study, an individual must meet all of the following criteria:

1. Age 1-65 years at the time of kidney transplant
2. Biopsy proven diagnosis of primary FSGS or minimal change disease
3. History of nephrotic syndrome (proteinuria, edema, hypoalbuminemia)
4. First kidney transplant or second or third transplant with a history of recurrent FSGS in the first or second kidney transplant.
5. The patient (if ≥18 years old) or the child's parent or guardian must be able and willing to give written informed consent and comply with the requirements of the study protocol. Patient assent if <18 years old will be required per local IRB requirements.
6. Negative urine pregnancy test prior to randomization (for females who are post-menarche).
7. Males and females of reproductive potential (sexually active in boys or post-menarche in girls) must agree to use an acceptable method of birth control during treatment and for twelve months (1 year) after completion of treatment with rituximab.

An individual who meets any of the following criteria will be excluded from participation in this study:

1. Known genetic cause of FSGS 2. Patients with FSGS secondary to another condition (obesity, viral infection, medications, etc.) 3. 4. Received rituximab within 1 year prior to transplant 5. Known hypersensitivity to rituximab, to any of its excipients, or to murine proteins 6. History of severe allergic or anaphylactic reactions to humanized or murine monoclonal antibodies 7. Known active bacterial, viral (e.g. HIV, hepatitis B, hepatitis C), fungal, mycobacterial, or other infection (including tuberculosis or atypical mycobacterial disease, but excluding fungal infections of nail beds) or any major episode of infection requiring hospitalization or treatment with iv antibiotics within 4 weeks of screening or oral antibiotics within 2 weeks prior to screening visit.

8. Participation in another therapeutic trial within 30 days of enrollment or 5 half-lives of the investigational drug (whichever is longer) 9. ANC < 1.5 x 103 10. Hemoglobin: < 8.0 gm/dL 11. Platelets: < 100,000/mm 12. AST or ALT >2.5 x Upper Limit of Normal at the local institution's laboratory 13. History of drug, alcohol, or chemical abuse within 6 months prior to screening visit.

14. Pregnant, lactating, or refusal of birth control in an adolescent of child-bearing potential 15. Concomitant malignancies or previous malignancies 16. History of psychiatric disorder that would interfere with normal participation in this protocol 17. History of significant cardiac (including arrhythmias) or pulmonary disease (including obstructive pulmonary disease) 18. Any other disease, metabolic dysfunction, physical examination finding, or clinical laboratory finding giving reasonable suspicion of a disease or condition that contraindicates the use of an investigational drug or that may affect the interpretation of the results or render the patient at high risk from treatment complications 19. Inability to comply with study and follow-up procedures

Ages: 1 Year to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 21 (Actual)
Dates: Start 2019-07-01 (Actual); Primary Completion 2025-02-07 (Actual); Study Completion 2025-02-07 (Actual)

PRIMARY OUTCOMES:
Feasibility assessment | through study completion, an average of 1 year
  quantifying the number and proportion of patients who can undergo the steps of recruitment, informed consent, enrollment, randomization, and follow-ups within the time frame of interest.

SECONDARY OUTCOMES:
Patient and graft survival at 1 year post-transplant | through study completion, an average of 1 year
  Outcome is reported as the number of participants who survive with a functional graft one year post-transplant.
Graft function at 1 year post-transplant | through study completion, an average of 1 year
  Graft function will be assessed using the glomerular filtration rate (GFR) and Schwartz equation (for age ≤17 years) or the CKD-EPI (for age ≥18 years).
Proportion with acute rejection at 1 year post-transplant | through study completion, an average of 1 year
  Outcome is reported as the percentage of participants who experience an acute graft rejection at one ear post-transplant.
Proportion with CD19+ <1% | 1 month, 6 months, and 12 months
  Outcome is reported as the percentage with participants with a reconstitution of CD19+ B cells at one year post-transplant.
Recurrent FSGS free survival | after 1 year post-transplant
  To determine the difference in rate of recurrent FSGS after 1 year post-transplant in patients receiving plasmapheresis and rituximab prior to or at the time of kidney transplantation compared to those receiving plasmapheresis alone.

CONTACTS AND LOCATIONS:
Overall Officials: Michelle Rheault, MD, Principal Investigator — University of Minnesota
Locations (12):
- United States (12):
  - University of Alabama, Tuscaloosa, Alabama
  - University of California at Davis, Davis, California
  - Lurie Children's Hospital, Chicago, Illinois
  - University of Iowa, Iowa City, Iowa
  - Children's Hospital of Colorado, Aurora, Minnesota
  - University of Minnesota, Minneapolis, Minnesota
  - Mayo Clinic, Rochester, Minnesota
  - Duke University, Durham, North Carolina
  - University of Cincinnati, Cincinnati, Ohio
  - Cincinnati Children's Hospital, Cincinnati, Ohio
  - Children's Hospital of Philadelphia, Philadelphia, Pennsylvania
  - Seattle Children's Hospital, Seattle, Washington

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Rheault MN, Amaral S, Bock M, Chambers ET, Chavers B, Ters ME, Garro R, Gbadegesin R, Govil A, Harshman L, Amer H, Hooper DK, Israni AK, Riad S, Sageshima J, Shapiro R, Seifert M, Smith J, Sung R, Thomas CP, Wang Q, Verghese PS. A randomized controlled trial of preemptive rituximab to prevent recurrent focal segmental glomerulosclerosis post-kidney transplant (PRI-VENT FSGS): protocol and study design. Front Nephrol. 2023 May 15;3:1181076. doi: 10.3389/fneph.2023.1181076. eCollection 2023. PMID 37675355